CLINICAL TRIAL: NCT00012428
Title: Prenatal PCB Exposure and Cognitive Development
Brief Title: Prenatal PCB Exposure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9815-CP-001
Record Dates: First submitted 2001-03-06; First posted 2001-03-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Maternal Exposure
Keywords: Cognitive development; Prenatal exposure; PCBs

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This project is designed to investigate the association between prenatal exposure to environmental contaminants on cognitive development of school-age children

ELIGIBILITY:
Pregnant mothers carrying full-term infants between 1991 and 1994. No longer recruiting. This is not a clinical trial. This is an epidemiological study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 224
Dates: Start 1999-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)